CLINICAL TRIAL: NCT02495831
Title: Drug Interaction Study of Safinamide and a BCRP Substrate, Diclofenac, Concomitantly Administered to Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zambon SpA (Industry)
Collaborators: Cross Research S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: Z7219J01
Record Dates: First submitted 2015-07-03; First posted 2015-07-13 (Estimated); Results first posted 2016-04-15 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Healthy
Keywords: PK study
MeSH Terms: interventions — Diclofenac; safinamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diclofenac sodium (Experimental): Diclofenac sodium 50 mg oral tablets, single dose
  Interventions: Drug: Diclofenac sodium
- Diclofenac sodium and safinamide (Active Comparator): Diclofenac sodium 50 mg oral tablets, single dose, and safinamide 200 mg oral tablets, single dose
  Interventions: Drug: Diclofenac sodium and safinamide

INTERVENTIONS:
Drug: Diclofenac sodium — Diclofenac sodium 50 mg single dose
  Other Names: Voltaren
  Arms: Diclofenac sodium
Drug: Diclofenac sodium and safinamide — Diclofenac 50 mg single dose and safinamide 200 mg single dose
  Other Names: Voltaren and Xadago
  Arms: Diclofenac sodium and safinamide

SUMMARY:
To evaluate if a single dose of safinamide 200 mg has an effect on the pharmacokinetics of diclofenamic acid, concomitantly administered as a single 50 mg diclofenac sodium dose, with respect to 50 mg diclofenac sodium administered alone.

DETAILED DESCRIPTION:
According to Xadago™ SmPC, safinamide may transiently inhibit BCRP, therefore a time interval of 5 h should be kept between dosing of safinamide and medicinal products that are BCRP substrates with a Tmax ≤2 h (e.g. diclofenac, pitavastatin, pravastatin, ciprofloxacin, methotrexate, topotecan or glyburide).

Following a specific request of EMA CHMP, the present interaction study in healthy male and female volunteers was conducted to determine if co-administration of safinamide with a BCRP substrate alters plasma exposure of the BCRP substrate in vivo.

Diclofenac was chosen among the other BCRP substrates considering its large use in the general population. Diclofenac in fact is an important analgesic and anti-inflammatory drug, widely used for the treatment of postoperative pain, rheumatoid arthritis, and chronic pain. Consequently, diclofenac is often used in combination regimens and undesirable drug-drug interactions may occur.

Voltaren®, 50 mg soluble tablets, was selected among other possible diclofenac products because with this formulation peak concentration of diclofenamic acid is achieved at approximately 1 h, i.e. in less than 2 h.

The present interaction study was designed in agreement with the FDA Guideline on Drug Interaction studies, taking also in consideration the EMA guideline on the Investigation of drug interactions.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent before inclusion in the study
2. Males and females, 25-55 years old
3. Body Mass Index (BMI): 18.5-30 kg/m2
4. Systolic blood pressure 100-139 mmHg, diastolic blood pressure 50-89 mmHg, heart rate 50-90 bpm
5. Ability to comprehend the full nature and purpose of the study
6. Females of child-bearing potential must use at least one of the following :

A non-hormonal intrauterine device or female condom with spermicide or contraceptive sponge with spermicide or diaphragm with spermicide or cervical cap with spermicide for at least 2 months before the screening visit A male sexual partner who agreed to use a male condom with spermicide A sterile sexual partner Female participants of non-child-bearing potential or in post-menopausal status for at least 1 year were admitted.

Exclusion Criteria:

1. Contraindications to MAO-B inhibitors, antiepileptic drugs, or to any NSAIDs
2. Clinically significant abnormalities in ECG
3. Clinically significant abnormal physical findings
4. Clinically significant abnormal laboratory values
5. Hypersensitivity or history of anaphylaxis to drugs or allergic reactions in general
6. Significant history of renal, hepatic, gastrointestinal, cardiovascular, respiratory, skin, haematological, endocrine or neurological diseases
7. Medications, including over the counter medications and herbal remedies, NSAID or anticoagulant use for 2 weeks before and during the entire study; morphine or other similar opioids, SSRIs, SNRIs, tri- or tetracyclic antidepressant, tramadol, pethidine, dextromethorphan, MAO inhibitors, meperidine derivatives and antiepileptic drugs, medicinal products that are BCRP substrates, any known enzyme inhibiting or inducing agent within 4 weeks preceding the screening visit.
8. Participation in the evaluation of any investigational product for 3 months before the study.
9. Blood donations for 3 months before the study
10. History of drug, alcohol, caffeine or tobacco abuse
11. Positive drug test at screening or day -1
12. Positive alcohol breath test at day -1
13. Abnormal diets or substantial changes in eating habits in the 4 weeks before the study; vegetarians
14. Positive or missing pregnancy test at screening or day -1, pregnant or lactating women

Ages: 22 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Milko Radicioni, MD, Principal Investigator — Cross Research SA
Locations (1):
- Cross Research SA, Phase I Unit, Arzo, Canton Ticino, Switzerland

IPD SHARING:
Plan to Share IPD: No
Bioequivalence data are to be considered as a whole in all subjects (90%CI).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment started and finished on May 2015 and the study was performed in Switzerland at CROSS Research S.A., Phase I Unit, Via F.A. Giorgioli 14 CH-6864 Arzo, Switzerland
Pre-assignment Details: Twenty-four (24) subjects were randomised in the study. One of the 24 subjects discontinued the study before study treatment. Twenty-two (22) subjects completed the study per protocol.
Groups:
- Diclofenac Sodium First, Safinamide + Diclofenac Sodium Second: Diclofenac sodium 50 mg oral tablets, single dose, and safinamide 200 mg oral tablets, single dose
- Safinamide + Diclofenac Sodium First, Diclofenac Sodium Second: Diclofenac sodium 50 mg oral tablets, single dose Safinamide 200 mg oral tablets, single dose
Period: First Intervention
Arm/Group | Diclofenac Sodium First, Safinamide + Diclofenac Sodium Second | Safinamide + Diclofenac Sodium First, Diclofenac Sodium Second
Started | 13 | 10
Completed | 13 | 10
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Diclofenac Sodium First, Safinamide + Diclofenac Sodium Second | Safinamide + Diclofenac Sodium First, Diclofenac Sodium Second
Started | 12 (One participant withdrew at the end of period 1) | 10
Completed | 12 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: males and females healthy volunteers, age 22-55 inclusive. This is a cross-over study, so 23 subjects were enrolled in total and participated in both groups
Groups:
- Intervention: Diclofenac sodium 50 mg oral tablets, single dose
  Diclofenac sodium 50 mg oral tablets, single dose and safinamide 200 mg oral tablets, single dose
Arm/Group | Intervention
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants] — healthy volunteers, both sexes, 22-55 years old inclusive
  Participants
    <=18 years | 0
    Between 18 and 65 years | 23
    >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.6 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Switzerland | 23

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate Plasma Diclofenamic Acid Extent of Exposure Reported as Plasma AUC After Single Administration of 50 mg Diclofenac Sodium, With and Without Co-administration of a Single 200 mg Dose of Safinamide.
Description: Plasma diclofenamic acid AUC0-t after T2 single dose, with and without T1 co-administration. To measure AUC plasma samples were taken by the participants at different time points, and the concentrations of diclofenac and safinamide were measured. AUC0-t is the area under the concentration-time curve from administration to the last observed concentration time t; PK parameters AUC0-t were analysed using analysis of variance (ANOVA). Before analysis, the data were transformed using a neperian logarithmic transformation. ANOVA was performed taking into account treatment, period, sequence and subject (sequence) as fixed effects with a variance components structure of the covariance matrix.
Time Frame: 24 hours
Population: healthy volunteers
Measure: Mean (Standard Deviation); unit: h X ng per mL
Arm/Group | Diclofenac Sodium | Diclofenac Sodium and Safinamide
Number analyzed (Participants) | 22 | 22
h X ng per mL | 1323.28 (390.53) | 1381.32 (393.77)
Statistical Analysis 1: Comparison: Diclofenac Sodium vs Diclofenac Sodium and Safinamide; The PK parameters AUC0-t and Cmax were analysed using analysis of variance (ANOVA). Before analysis, the data were transformed using a neperian logarithmic transformation. ANOVA was performed taking into account treatment, period, sequence and subject (sequence) as fixed effects with a variance components structure of the covariance matrix; Test type: Superiority or Other; p = 0.1, ANOVA — If the upper limit of the 90% confidence interval is < 125.00%, no effect of safinamide on diclofenamic acid bioavailability is present (no interaction present); point estimate (ratio of geometric means = 90, 90% CI 2-sided [80 to 125]

2. Secondary Outcome: Evaluate Diclofenac Rate of Absorption Reported as Plasma Cmax After Single Administration of 50 mg Diclofenac With and Without 200 mg of Safinamide.
Description: Cmax, of plasma diclofenamic acid after T2 single dose, with and without T1 co-administration. The parametric point estimators (PE) for the ratios of T2 treatment with T1 co-administration / T2 treatment without T1 co-administration for the PK parameters under consideration, and the two-sided 90% confidence interval (CI), were calculated using the adjusted least squares means (LSMEANS) from the ANOVA. LSmeans differences obtained in the log scale for Cmax were back-transformed to obtain the PE (i.e. geometric mean ratio) and the two-sided 90% CI as percentages.
Time Frame: 24 hours
Measure: Least Squares Mean (Standard Deviation); unit: ng/mL
Arm/Group | Diclofenac Sodium | Diclofenac Sodium and Safinamide
Number analyzed (Participants) | 22 | 22
ng/mL | 766.59 (390.01) | 833.50 (443.34)
Statistical Analysis 1: Comparison: Diclofenac Sodium vs Diclofenac Sodium and Safinamide; Test type: Superiority or Other; geometric mean ratio = 104.84, 90% CI 2-sided [96.40 to 114.02]

3. Secondary Outcome: Tmax and T1/2
Time Frame: 24 hours
Measure: Least Squares Mean (Standard Deviation); unit: hours
Arm/Group | Diclofenac Sodium | Diclofenac Sodium and Safinamide
Number analyzed (Participants) | 22 | 22
hours
  Tmax | 0.88 (0.41) | 1.0 (0.43)
  T1/2 | 1.24 (0.43) | 1.19 (0.40)

4. Secondary Outcome: Lamda z
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: 1/hours
Arm/Group | Diclofenac Sodium | Diclofenac Sodium and Safinamide
Number analyzed (Participants) | 22 | 22
1/hours | 0.63 (0.22) | 0.63 (0.16)

5. Secondary Outcome: Relative Bioavailability (Frel)
Description: calculated as ratio between AUC0-t (test) / AUC0-t (reference)
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Diclofenac Sodium | Diclofenac Sodium and Safinamide
Number analyzed (Participants) | 22 | 22
ratio | 107.67 (28.84) | 109.61 (32.14)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Diclofenac Sodium | Diclofenac Sodium and Safinamide
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23

LIMITATIONS AND CAVEATS:
no limitations

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less